CLINICAL TRIAL: NCT02485509
Title: Phase Ib/IIa, Single-Centre, Placebo-Controlled Randomized Study of Safety and Pharmacokinetics in Healthy Volunteers and Safety, Tolerability and Antiviral Activity of VM-1500 in Patients With Human Immunodeficiency Virus-1 Infection
Brief Title: Study of Safety and Pharmacokinetics in Healthy Volunteers and Safety, Tolerability and Antiviral Activity of VM-1500 in Patients With Human Immunodeficiency Virus-1 Infection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Viriom (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VM-1500-001
Record Dates: First submitted 2015-06-18; First posted 2015-06-30 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 20 mg VM-1500/Placebo Healthy group (Experimental): VM-1500 20 mg or placebo single dose.
  Interventions: Drug: VM-1500/Placebo
- 40 mg VM-1500/Placebo Healthy group (Experimental): VM-1500 40 mg or placebo single dose.
  Interventions: Drug: VM-1500/Placebo
- 20 mg VM-1500/Placebo Patient group (Experimental): VM-1500 20 mg or placebo once daily for 7 days.
  Interventions: Drug: VM-1500/Placebo
- 40 mg VM-1500/Placebo Patient group (Experimental): VM-1500 40 mg or placebo once daily for 7 days.
  Interventions: Drug: VM-1500/Placebo

INTERVENTIONS:
Drug: VM-1500/Placebo — VM-1500 or Placebo

SUMMARY:
A combined Phase Ib and IIa randomized, placebo-controlled, double-blind study of VM-1500 in healthy subjects and in patients with HIV-1 infection that are antiretroviral therapy naïve.

DETAILED DESCRIPTION:
The study will be split into two parts:

Part I: A randomized, placebo-controlled, single dose, double-blind study in healthy volunteers with 20 mg followed by 40 mg after DSMB approval.

Healthy group: one dose with 1 PK day 12 health volunteers (total): 6 subjects will randomized (4:2) to VM-1500 20 mg or placebo. After DSMB approval, 6 subjects will be randomized (4:2) to VM-1500 40 mg or placebo Part II: A randomized, placebo-controlled, multiple dose, double-blind study for 7 days in patients with HIV infection who are antiretroviral therapy-naïve. After positive DMSB review the dose will be escalated from 20 mg to 40 mg once daily.

Patient group: 2 PK days (in-house) at day 1 and day 7 16 patients (total): 8 subjects will be randomized (7:1) to VM-1500 20 mg or placebo once daily for 7 days. After DSMB approval, 8 subjects will be randomized (7:1) to VM-1500 40 mg or placebo once daily for 7 days.

ELIGIBILITY:
Inclusion Criteria for Healthy Subjects:

1. Male age between 18-40 years
2. Has been determined healthy by physical examination, assessment of drug abuse, medical history and vital signs
3. Has normal results for the following screening tests: complete blood count , blood urea nitrogen, serum creatinine , fasting blood sugar, total bilirubin, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase and urinalysis.
4. Negative result for hepatitis B, hepatitis C and HIV antibodies
5. Willing to participate and signed the informed consent form

   Inclusion Criteria for Patients:
6. Males or females aged 18 to 65 years
7. HIV-1 infection, as documented by a rapid HIV test or any licensed ELISA test kit and confirmed by Western blot at any time prior to study entry
8. Antiretroviral therapy naïve.

Exclusion Criteria for Healthy Subjects:

1. Hepatic or kidney disorders or any other disease or disorder which may in the opinion of the Investigator interfere with the results of the study or threaten the health of volunteers;
2. Drug intake (including herbal drugs) during the last month;
3. Active alcohol or and/or drug abuse that, in the opinion of the site investigator, would interfere with adherence to study requirements;
4. Volunteers have taken any investigational drug at least 3 month prior to the start of the study;
5. Inability to understand the Protocol or follow its instructions;

Exclusion Criteria for Patients:

1. Currently has any active AIDS defining illness
2. Exclusionary resistance mutations defined as evidence of any major NNRTI mutations according to the current IAS list of HIV-1 Resistance Mutations Associated with Drug Resistance on any genotype; or evidence of significant NNRTI resistance on any phenotype performed at any time prior to study entry.
3. Patients who are expected to need systemic antiviral therapy at any time during their participation in the study.
4. Patients who have received an investigational drug for HIV, HIV vaccine, immunomodulators, systemic cytotoxic chemotherapy, or other investigational therapy within 30 days prior to study entry;
5. Acute or chronic viral hepatitis;
6. History or other evidence of renal disease.
7. Abnormal hematological and biochemical parameters within 30 days of Entry (Day 1).
8. Screening ECG QTc value 450 ms.
9. Consumption / administration of concomitant medication.
10. Active alcohol and/or drug abuse that, in the opinion of the site investigator, would interfere with adherence to study requirements.
11. Positive results on urine screen for drugs of abuse at Screening or Day 1
12. History of immunologically mediated disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of VM-1500 in adult healthy subjects and in patients with early-stage chronic HIV-1 infection based on analysis of AEs, laboratory values. | about one and half month

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile of VM-1500 in healthy subjects (Cmax, AUC, T1/2) and in HIV-1-infected patients. | about one and half month
Dose dependency between VM-1500 plasma levels and corresponding HIV RNA reduction with the administered dosages of VM-1500. | about one and half month
Virologic activity as measured by plasma HIV RNA following treatment for seven (7) days with VM-1500. | about one and half month

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Siriraj Hospital, Bangkok, Wanglang Road, Thailand